CLINICAL TRIAL: NCT04805632
Title: A Comparison of Short-term and Mid-term Immune Response in Dialysis Patients and Staff Vaccinated Against SARS-CoV-2 Using Gam-COVID-Vac (Sputnik V) Vaccine
Brief Title: Immune Response in Dialysis Patients Vaccinated Against COVID-19
Acronym: Sputnik-HD
Status: Completed | Type: Observational
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Ekaterina Parshina, Principal investigator, MD, Saint Petersburg State University, Russia
Other Study IDs: Sputnik_HD
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Covid19; Chronic Kidney Disease 5D
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dialysis: Patients on hemodialysis or peritoneal dialysis who received 2 administrations of Gam-COVID-Vac (Sputnik V) vaccine against SARS-CoV-2 infection
- Healthy: Medical staff who received 2 administrations of Gam-COVID-Vac (Sputnik V) vaccine against SARS-CoV-2 infection

SUMMARY:
This is a prospective cohort study aimed to evaluate short- and mid-term immune response after SARS-CoV-2 vaccination using Gam-COVID-Vac (Sputnik V) vaccine in dialysis patients compared to the control group (medical staff).

DETAILED DESCRIPTION:
Background and aims: Patients receiving kidney replacement therapy with dialysis are at high risk of infection and death from COVID-19. There is a lack of evidence whether SARS-CoV-2 vaccination is effective in this immunocompromised group.

Study design: this is a prospective cohort study. Two cohorts will be included: dialysis patients and controls (medical staff), both vaccinated with Gam-COVID-Vac (Sputnik V) vaccine.

Blood samples will be collected at 28 days and 22 weeks after after the second SARS-CoV-2 vaccine dose administration.

The primary outcome is the level of SARS-CoV-2 IgG antibodies on day 28 after the second vaccination as compared to controls.

The secondary outcomes are: 1) the level of SARS-CoV-2 IgG antibodies on week 22 after the second vaccination; 2) T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) 28 days and 22 weeks after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Previously vaccinated against SARS-CoV-2 with two administrations of Gam-COVID-Vac (Sputnik V) vaccine
* Written informed consent.

Exclusion Criteria:

* A history of previous COVID-19 disease
* Active malignancy of any localization
* Human Immunodeficiency Virus (HIV) infection
* Maintenance treatment with immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years old who were vaccinated twice against SARS-CoV-2 using Gam-COVID-Vac (Sputnik V) vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Humoral response to vaccination against against SARS-CoV-2 as compared to controls | 28 days after the second vaccination
  SARS-CoV2 IgG levels

SECONDARY OUTCOMES:
Humoral response to vaccination against against SARS-CoV-2 | 22 weeks after the second vaccination
  SARS-CoV2 IgG levels
T-cell response against SARS-CoV-2 | 28 days after the second vaccination
  SARS-CoV-2 specific T-cell subtype measured by interferon-γ release assays (IGRA)
T-cell response against SARS-CoV-2 | 22 weeks after the second vaccination
  SARS-CoV-2 specific T-cell subtype measured by interferon-γ release assays (IGRA)
SARS-CoV-2 incidence | 22 weeks after the second vaccination
  Survey of the incidence of SARS-CoV-2 infections over the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia